CLINICAL TRIAL: NCT05282303
Title: REGIONAL ANALGESIA TECHNIQUES FOR EFFECTIVE RECOVERY TO CORONARY ARTERY BYPASS SURGERIES: A RETROSPECTİVE STUDY IN A SINGLE CENTER EXPERIENCE
Status: Completed | Type: Observational
Sponsor: V.K.V. American Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Sami Kaan Coşarcan, MD, V.K.V. American Hospital, Istanbul
Other Study IDs: Cosarcan3
Record Dates: First submitted 2022-02-25; First posted 2022-03-16 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- DIESPB: Dual injection of erector spinae plane block
  Interventions: Procedure: CABG operation
- TPVB: Thoracic paravertebral block
  Interventions: Procedure: CABG operation
- SAB: Serratus anterior plane block
  Interventions: Procedure: CABG operation
- PIB: Parasternal ıntercostal block
  Interventions: Procedure: CABG operation

INTERVENTIONS:
Procedure: CABG operation — Efficacy of regional analgesia techniques in coronary artery bypass operations

SUMMARY:
Background Pain after cardiac surgery is both multifocal and multifactorial. Sternotomy, sternal retraction, internal mammary dissection, posterior rib dislocation or fracture, possible brachial plexus injury, and mediastinal and pleural drains contribute to pain experienced in the immediate postoperative period. Ineffective pain management can cause systemic and pulmonary complications and significant cardiac consequences.

Methods This study was conducted to compare the effectiveness of regional anesthesia techniques for perioperative pain management in cardiac surgery patients at our clinic. The effects of analgesic methods, in terms of contributing to recovery, have been examined.

DETAILED DESCRIPTION:
This study was approved by the Koç University Clinical Research Ethics Committee (2021.464.IRB1.131); patients who underwent coronary artery bypass grafting (CABG) surgery at the VKV American Hospital between January 2015 and May 2020 were reviewed retrospectively. Patients with a history of cerebrovascular events, scheduled carotid surgery, or emergency CABG surgery were excluded from the study. Demographic data from the preoperative evaluation forms and operation types from the surgery reports were recorded. Intraoperative anesthesia follow-up forms were assessed if regional anesthesia was used, and the type and extent of opioids during the operation were examined. The postoperative transfer forms were examined to the cardiovascular intensive care unit (CICU), intensive care follow-up forms, and service ward record follow-up forms. Pain scores (NRS) during rest and coughing, vital signs, mobilization, and the start of respiratory exercises were recorded for postoperative respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* Who underwent coronary artery bypass grafting (CABG) surgery at the VKV American Hospital between January 2015 and May 2020 were reviewed retrospectively

Exclusion Criteria:

* History of cerebrovascular event
* History of Alzheimer's and dementia
* Inadequate cognitive functions
* History of chronic pain
* Long-term opioid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease scheduled for bypass surgery
Sampling Method: Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
Postoperative analgesia | 0 - 24 hours
  NRS score

CONTACTS AND LOCATIONS:
Locations (1):
- American Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Bigeleisen PE, Goehner N. Novel approaches in pain management in cardiac surgery. Curr Opin Anaesthesiol. 2015 Feb;28(1):89-94. doi: 10.1097/ACO.0000000000000147. PMID 25500688
- [Result] Doehring A, Oertel BG, Sittl R, Lotsch J. Chronic opioid use is associated with increased DNA methylation correlating with increased clinical pain. Pain. 2013 Jan;154(1):15-23. doi: 10.1016/j.pain.2012.06.011. PMID 23273101
- [Result] Nagaraja PS, Ragavendran S, Singh NG, Asai O, Bhavya G, Manjunath N, Rajesh K. Comparison of continuous thoracic epidural analgesia with bilateral erector spinae plane block for perioperative pain management in cardiac surgery. Ann Card Anaesth. 2018 Jul-Sep;21(3):323-327. doi: 10.4103/aca.ACA_16_18. PMID 30052229
- [Result] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Result] Elsharkawy H, Pawa A, Mariano ER. Interfascial Plane Blocks: Back to Basics. Reg Anesth Pain Med. 2018 May;43(4):341-346. doi: 10.1097/AAP.0000000000000750. PMID 29561295